CLINICAL TRIAL: NCT01108835
Title: A Comprehensive Care Programme for Patients With Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Fanny W.S. Ko, Honorary Associate Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Resp/Ko/2010/001
Record Dates: First submitted 2010-04-16; First posted 2010-04-22 (Estimated); Results first posted 2017-03-30 (Actual); Last update posted 2017-08-23 (Actual); Status verified 2017-07

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; Comprehensive care
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- comprehensive care programme (Active Comparator): Comprehensive care involving multidisciplinary input.
  Interventions: Other: Comprehensive care programme
- Control group (No Intervention): Control arm with usual care

INTERVENTIONS:
Other: Comprehensive care programme — Intervention group:
  * Patients will be interviewed by a respiratory nurse and given education in 1-2 sessions
  * Physiotherapist assessment and training (individualized physical training programme to perform at home or a short course out-patient pulmonary rehabilitation)
  * Respiratory physician assessment and optimization of treatment
  * Patients will also be taught about a personalized action plan by the physician and respiratory nurse.
  * Subsequent intervention: Patients will receive monthly telephone calls by a respiratory nurse for a period of 1 year to assess their conditions and also answer their queries.
  Arms: comprehensive care programme

SUMMARY:
Objective: Chronic obstructive pulmonary disease (COPD) is a disease with significant morbidity and incurs heavy utilization of healthcare resources. The direct cost of hospital admissions related to COPD is the single largest source of expenditure in the public hospital system. This study aims to assess whether a comprehensive care programme can decrease the rate of hospital admissions for COPD patients.

DETAILED DESCRIPTION:
Design: A randomised controlled trial of patients discharged from hospital after an episode of acute exacerbation of COPD. Patients will be randomised to the intervention arm or usual care group.

Setting: Tertiary University affiliated Hospital.

Interventions:

The Intervention group will receive a comprehensive programme which involves inputs from doctors, respiratory nurses and physiotherapists, providing an individualized care plan for each subject. The components in the programme will include optimization of medications, specialist physician follow up, nursing support in education, and physiotherapist support for pulmonary rehabilitation. Patients in the intervention group will also receive monthly telephone calls by a respiratory nurse for a period of 1 year to assess their conditions and answer their queries. Patients will also be followed up in the respiratory clinic by respiratory specialist once every 3 months for 1 year.

The control group will be managed as the usual care. The discharging physician will determine the patients' medication and follow up as in normal practice.

All patients will be asked to return for assessments (spirometry, 6 minute walk test, questionnaires on the severity of dyspnoea and quality of life) at baseline and 12 months

Main outcome measures: The primary endpoint is the hospital readmission rate and the secondary endpoints are the quality of life, mortality, lung function and exercise capacity of the patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are admitted to the Prince of Wales Hospital with AECOPD will be screened for this study.
* Patients with age over 40 years

Exclusion Criteria:

* Patients with asthma
* Patients unable to provide informed consent

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2010-04; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David S Hui, MD, Study Director — Chinese University of Hong Kong
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ko FW, Cheung NK, Rainer TH, Lum C, Wong I, Hui DS. Comprehensive care programme for patients with chronic obstructive pulmonary disease: a randomised controlled trial. Thorax. 2017 Feb;72(2):122-128. doi: 10.1136/thoraxjnl-2016-208396. Epub 2016 Jul 28. PMID 27471050

RESULTS

PARTICIPANT FLOW:
Groups:
- Comprehensive Care: Comprehensive care
  Comprehensive care programme: Intervention group:
  * Patients will be interviewed by a respiratory nurse and given education in 1-2 sessions
  * Physiotherapist assessment and training (individualized physical training programme to perform at home or a short course out-patient pulmonary rehabilitation)
  * Respiratory physician assessment and optimization of treatment
  * Patients will also be taught about a personalized action plan by the physician and respiratory nurse.
  * Subsequent intervention: Patients will receive monthly telephone calls by a respiratory nurse for a period of 1 year to assess their conditions and also answer their queries.
Period: Overall Study
Arm/Group | Comprehensive Care | Control Group
Started | 90 | 90
Completed | 73 | 69
Not Completed | 17 | 21

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Comprehensive Care | Control Group | Total
Number analyzed (Participants) | 90 | 90 | 180
Age, Customized [Mean (Standard Deviation); unit: years]
  Age (years) | 74.9 (7.9) | 74.6 (8.6) | 74.7 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 8
  Male | 85 | 87 | 172
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 90 | 90 | 180
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants] — All subjects are recruited from Hong Kong.
  participants
    Hong Kong | 90 | 90 | 180

OUTCOME MEASURES:

1. Primary Outcome: Hospital Readmission
Description: To investigate the effectiveness of a comprehensive care programme in reducing hospital admission in COPD patients who have been discharged from hospital for an episode of AECOPD.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: hospital readmissions
Arm/Group | Comprehensive Care | Control Group
Number analyzed (Participants) | 90 | 90
hospital readmissions | 1.12 (1.69) | 1.7 (1.65)

2. Secondary Outcome: Quality of Life
Description: Measured by change in St. George Respiratory Questionnaire (SGRQ) total score from baseline to 12 month. SGRQ total score ranged from 0-100. The change was calculated by the 12 month SGRQ total score minus the baseline value. Negative values indicated improvement in quality of life.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Comprehensive Care Programme: Comprehensive care involving multidisciplinary input.
  Comprehensive care programme: Intervention group:
  * Patients will be interviewed by a respiratory nurse and given education in 1-2 sessions
  * Physiotherapist assessment and training (individualized physical training programme to perform at home or a short course out-patient pulmonary rehabilitation)
  * Respiratory physician assessment and optimization of treatment
  * Patients will also be taught about a personalized action plan by the physician and respiratory nurse.
  * Subsequent intervention: Patients will receive monthly telephone calls by a respiratory nurse for a period of 1 year to assess their conditions and also answer their queries.
Arm/Group | Comprehensive Care Programme | Control Group
Number analyzed (Participants) | 90 | 90
units on a scale | -6.9 (15.3) | -0.1 (15.7)

3. Secondary Outcome: Mortality
Description: From contacting the patient/their family and hospital record retrieval.
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | Comprehensive Care | Control Group
Number analyzed (Participants) | 90 | 90
participants | 10 | 12

4. Secondary Outcome: Lung Function
Description: Measurement of change of spirometry (FEV1 % predicted) from baseline to 12 month. The range is from 0% to 100%. The change was calculated by 12 month value minus the baseline value. Positive value indicated improvement in lung function.
Time Frame: 12 months
Population: Percentage of predicted FEV1
Measure: Mean (Standard Deviation); unit: Percentage of Predicted FEV1
Arm/Group | Comprehensive Care | Control Group
Number analyzed (Participants) | 90 | 90
Percentage of Predicted FEV1 | 0.8 (6.8) | -0.5 (8.5)

5. Secondary Outcome: Exercise Capacity
Description: Exercise capacity was measured by change in 6 minutes walk test distance from baseline to 12 month. 6 minute walk test is the distance that the patient can walk over 6 minutes and it can range to 0 meters to few hundred meters. This was calculated by the 12 month 6 minutes walk test distance minus that of the baseline. Positive values indicated improvement in exercise capacity.
Time Frame: 12 month
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Comprehensive Care | Control Group
Number analyzed (Participants) | 90 | 90
meters | -10.0 (61.2) | -22.5 (71.4)

ADVERSE EVENTS:
Time Frame: 12 months
Description: adverse events
Arm/Group | Comprehensive Care | Control Group
Serious Adverse Events (participants affected / at risk) | 0/90 | 0/90
Other Adverse Events (participants affected / at risk) | 0/90 | 0/90

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No